CLINICAL TRIAL: NCT02651961
Title: Cost-effectiveness Evaluation of One Stage Versus Two Stage Exchange for Chronically Infected Total Hip and Total Knee Prostheses
Acronym: IPRO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 6262
Record Dates: First submitted 2015-11-25; First posted 2016-01-11 (Estimated); Last update posted 2018-05-22 (Actual); Status verified 2018-05

CONDITIONS: Chronically Infected Total Hip of Knee Prosthesis
Keywords: Total hip prosthesis; Total knee prosthesis; Chronic infection; One stage exchange; Two stage exchange; Cost-effectiveness
MeSH Terms: conditions — Persistent Infection | interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- One stage exchange (Active Comparator): One stage exchange of the chronically infected implant
  Interventions: Procedure: Exchange of total hip or knee arthroplasty on same time
- Two stage exchange (Active Comparator): Two stage exchange of the chronically infected implant
  Interventions: Procedure: Exchange of total hip or knee arthroplasty in two time

INTERVENTIONS:
Procedure: Exchange of total hip or knee arthroplasty on same time — Removal of the index implants, extensive debridement, reimplantation of a new prosthesis
  Arms: One stage exchange
Procedure: Exchange of total hip or knee arthroplasty in two time — Removal of the index implants in first time, extensive debridement, reimplantation of a new prosthesis in seconde time
  Arms: Two stage exchange

SUMMARY:
Chronic infection after total joint arthroplasty generally requires implant exchange. Two stage exchange is considered as the gold standard procedure. However, some authors suggest that one stage exchange may be as effective. No consensus exists in the current literature. The purpose of the study was to evaluate the cost of both strategies in comparison to their success rate.

DETAILED DESCRIPTION:
The primary criterion will be the cost-utility ratio (ICER) at 12 months follow-up.

The secondary criteria will be:

* quality of life;
* pain;
* persistence or recurrence of infection;
* occurrence of complications ;
* necessity for reoperation.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Chronically infected total hip or knee arthroplasty requiring implant exchange
* Affiliation to a social security system
* Signed informed consent
* Effective contraception during all study

Exclusion Criteria:

* Repeat exchange after failure of a prior treatment for infection
* Multiple implant infection
* Infection due to mycobacteria or fungus
* Pregnancy / Breast feeding
* Patient under judicial protection
* Impossibility to give informed consent for any reason
* Participation to another study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-05-03 (Actual); Primary Completion 2022-10-02 (Estimated); Study Completion 2022-10-02 (Estimated)

PRIMARY OUTCOMES:
Cost-utility ratio (ICER) | 12 months post-operative

SECONDARY OUTCOMES:
Quality of life : EQ-5D questionnaire | 12 months post-operative
  Patient-reported generic (EQ-5D) outcomes questionnaire
Pain : VAS score | 12 months post-operative
  Patient-reported pain score with visual analogic scale
Number of Persistence or recurrence of infection for all participants | 24 months post-operative
Occurrence of complications | 24 months post-operative
number of Necessity of reoperation for all patient | 12 months post-operative
  necessity of reoperation will be assessed with clinical examination
Operating time of all surgical procedures | procedure
  operating time is from time of entrance in the operating room to time of the end of intervention (hh:mm)
Duration of whole treatment | 12 months post-operative
Cost of complication treatment | 12 months post-operative
Cost of repeat surgery | 12 months post-operative
Quality of life : Oxford hip or knee questionnaires | 12 months post-operative
  Patient-reported specific (Oxford) outcomes questionnaire
cost of whole treatment | 12 months post-operative

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Yves JENNY, PH, Principal Investigator — Strasbourg's University Hospitals
Locations (1):
- Hôpitaux Universitaires de Strasbourg, Strasbourg, France